CLINICAL TRIAL: NCT00446303
Title: A Phase II Study of Maintenance With Azacitidine in MDS Patients Achieving Complete or Partial Remission (CR or PR) After Intensive Chemotherapy
Brief Title: A Phase II Study of Maintenance With Azacitidine in MDS Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GFM aza05
Record Dates: First submitted 2007-03-09; First posted 2007-03-12 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2010-06

CONDITIONS: Leukemia, Myelocytic, Acute; Myelodysplastic Syndromes
Keywords: MDS; Myelodysplastic Syndromes; AML; Intensive chemotherapy; azacitidine
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Azacitidine — Azacitidine 60mg/m2 /d for 5 days every 28 days, for 24 months (parallel study to the ongoing NMDSG study.
  Extension of maintenance in responders after 24 courses until relapse or death.

SUMMARY:
A phase II multicentre trial of maintenance with Azacitidine in MDS patients achieving complete or partial remission (CR or PR) after intensive chemoterapy.

The primary objective is response duration (MDS or AML)

DETAILED DESCRIPTION:
A academic multicentre study whose aims are to study the benefits of a maintenance therapy with 24 monthly courses af azacytidine in high-risk MDS patients, previously treated with intensive chemotherapy with obtention of a partial or complete response and not eligible for allogeneic transplantation

ELIGIBILITY:
Inclusion Criteria:

* MDS with int 2 or high IPSS score eitherRAEB 1 or 2 according to the WHO classification (see appendix 1) or CMML with WBC < 13 109/l RAEB-T according to the FAB classification (see appendix 1) without t(8 ;21), inv 16 or t(16;16) AML secondary to MDS (sAML) with a confirmed MDS phase of at least 2 months with available bone marrow cytogenetics at diagnosis of AML

AND

in CR or PR according to IWG criteria (see appendix 3) after one or two courses of predefined intensive chemotherapy (see page 12) with available cytogenetics at evaluation of response Aged 18 years of age or more Written Informed consent Adequate Contraception, if relevant Negative pregnancy test if relevant. Patients not eligible for the azacitidine confirmatory trial (azacitidine " versus " conventional treatment ") or unwilling to participate to it

Exclusion Criteria:

* AML secondary to myeloproliferative or MDS/MPD WHO subgroups except CMML with WBC< 13 109/l
* Therapy related MDS (after chemo or radiotherapy for a previous neoplasm or immune disorder)
* Patients eligible for allogeneic bone marrow transplantation (with a identified donor)
* Liver and/or kidney failures prohibiting the use of azacitidine. Creatininemia > 1.5 normal value ALAT and ASAT > 3N
* Bilirubin > 2 N, unless due to dyserythropoiesis
* Known hypersensitivity to azacitidine or mannitol
* Other tumor, unstable for the last three years, except in situ uterine carcinoma or basal skin tumor
* Uncontrolled infection,
* WHO Performance status > 2
* Life expectancy less than 3 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2006-07; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Reponse duration and cumulative incidence of relapses | 1-24 months

SECONDARY OUTCOMES:
Toxicity according to WHO | 1-24 months
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Claude GARDIN, MD, Principal Investigator — Groupe Francophone des Myelodysplasies
Locations (25):
- France (25):
  - CHU d'Amiens, Amiens
  - CHU Angers, Angers
  - CH d'Avignon, Avignon
  - CHU de Caen, Caen
  - Hopital d'Instruction des Armées Percy, Clamart
  - Hopital Henri Mondor, Créteil
  - CHU de Dijon, Dijon
  - CHU Albert Michallon, Grenoble
  - CHRU Hurriez, Lille
  - CHRU de Limoges, Limoges
  - Hopital Edouard Herriot, Lyon
  - Hopital Paoli Calmette, Marseille
  - Hopital Hotel Dieu, Nantes
  - Hopital Archet, Nice
  - Hopital Saint Louis, Paris
  - Hopital Saint Antoine, Paris
  - Hopital Cochin, Paris
  - Hopital Haut Leveque, Pessac
  - Hopital Jean-Bernard, Poitiers
  - CHRU de Reims, Reims
  - CHU Pontchaillou, Rennes
  - Hopital Hautepierre, Strasbourg
  - Hopital Purpan, Toulouse
  - CHU Brabois, Vandœuvre-lès-Nancy
  - CH Versailles, Versailles